CLINICAL TRIAL: NCT05811780
Title: The University of Freiburg Medical Center Extracorporeal Organ Support Device Registry
Status: Recruiting | Type: Observational
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, PD Dr. Alexander Supady, Co-Principal Investigator, University Hospital Freiburg
Other Study IDs: 151/14
Record Dates: First submitted 2023-03-20; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Medical Condition Requiring Extracorporeal Organ Support
Keywords: Acute Respiratory Distress Syndrome; acute respiratory failure; severe respiratory failure; cardiogenic shock; cardiac arrest; extracorporeal cardiopulmonary resuscitation
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Insufficiency; Shock, Cardiogenic; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective registry collecting pseudonymized clinical and treatment data from all patients treated with extracorporeal organ support (i.e., VV ECMO, VA ECMO, ECPR, Impella, IABP, and others) on the wards of the Department of Interdisciplinary Medical Intensive Care at the Freiburg University Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with any kind of extracorporeal organ support

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients receiving extracorporeal organ support and being treated in the Department of Interdisciplinary Medical Intensive Care of the Freiburg University Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2014-04-29 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospital survival | 30 days
  Survival of index hospitalization (yes/no)

OTHER OUTCOMES:
Mesenteric ischemia | 30 days
  Occurrence of mesenteric ischemia
Fluid balance | 7 days
  Patient fluid balance (difference between fluid input and output)
ECMO run-time | 60 days
  Duration of ECMO support

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Wengenmayer, Prof. Dr., Study Director — University of Freiburg; Dawid L Staudacher, PD Dr., Principal Investigator — University of Freiburg; Paul M Biever, Dr., Principal Investigator — University of Freiburg; Jonathan Rilinger, PD Dr., Principal Investigator — University of Freiburg; Alexander Supady, PD Dr., Principal Investigator — University of Freiburg
Locations (1):
- University of Freiburg Medical Center, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No